CLINICAL TRIAL: NCT05715710
Title: Correlation Between Deep Medullary Veins and Cognitive Dysfunction in Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: Zigong No.1 Peoples Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022ZCNKY08
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Small Vessel Disease
Keywords: deep medullary veins; csvd; cerebral small vessel disease
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to obtain the characteristics of cognitive impairment and imaging characteristics of patients with Cerebral small vessel disease (CSVD) through comprehensive and standardized neuropsychological assessment and multimodal imaging examination. The focus is to obtain the characteristics of cognitive impairment and imaging characteristics of patients with CSVD through 3.0T MRI SWI sequence. deep medullary veins (DMVs) were measured. To compare the demographic data, hematological indexes, imaging scores and the number of DMVs between CSVD groups with and without cognitive impairment, and to explore the correlation between deep medullary veins and cognitive dysfunction in cerebral small vessel disease.

DETAILED DESCRIPTION:
This study aims to obtain the characteristics of cognitive impairment and imaging characteristics of patients with Cerebral small vessel disease (CSVD) by conducting comprehensive and standardized neuropsychological assessment and multimodal imaging examination. deep medullary veins (DMVs) were measured. The demographic data, hematological indexes, imaging scores and the number of DMVs were compared between the CSVD group with and without cognitive impairment, and the risk factors for cognitive impairment in CSVD were analyzed to explore whether DMVs could be an independent risk factor for cognitive impairment in CSVD. To establish a multiple model for the risk prediction of cognitive impairment in CSVD, and to understand whether the prediction model combined with the number of DMVs has a better prediction effect on cognitive impairment in CSVD. In order to find new imaging markers of cognitive impairment in CSVD, and provide evidence for early detection and intervention of cognitive impairment in clinical CSVD.

ELIGIBILITY:
1. Inclusion Criteria

   1. Age 50 ~ 85 years old.
   2. The diagnostic criteria of CSVD patients with cerebral small vessel diseases should be in accordance with the 2015 Chinese Consensus on the diagnosis and treatment of cerebral small vessel Diseases formulated and recommended by the Cerebrovascular Division of Chinese Society of Neurology, Chinese Medical Association. MRI examination revealed the presence of one or more of the major imaging features of CSVD as proposed by the 2013 International Standards Reporting Group on Neuroimaging of Vascular Changes.
   3. No large vessel stenosis (stenosis rate > 50%) was found after head and neck vascular examination (CTA, MRA, DSA or TCD combined with carotid ultrasound).
   4. The vital signs are stable and can cooperate with the examination.
   5. Informed consent signed by the patient or legal representative.
2. Exclusion Criteria:

   1. Cerebral infarction or cerebral hemorrhage caused by large vascular disease; And CTA/MRA of the head and neck showed great vessel stenosis (stenosis rate > 50%).
   2. Patients with secondary white matter lesions caused by poisoning, inflammation, tumor and other pathological changes.
   3. Cognitive impairment and gait impairment caused by other causes (such as Alzheimer's disease, Parkinson's disease, depression, etc.
   4. Patients with contraindications of magnetic resonance examination.
   5. Illiterate or unable to cooperate with cognitive assessment due to severe hearing and visual impairment.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. CSVD patients who met the inclusion and exclusion criteria were included. Demographic data, cerebrovascular disease risk factors data, and hematological data were collected.
  2. Standardized neuropsychological assessment was performed to evaluate the general cognition and various cognitive domains (memory, language, visuospatial execution) of CSVD patients.
  3. Fazekas score of white matter hyperintensity (WMH) and cerebral microbleed (cerebral microbleed) were calculated based on the results of 3.0 T multimode MRI examination. CMB count, lacunar infarction count, perivascular space (PVS) count, and MRI total load score; Deep medullary veins (DMVs) were counted by SWI sequence.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Deep medullary veins score | 2022.01-2025.1
  In this study, deep medullary veins (DMVs) were counted by SWI sequence.

CONTACTS AND LOCATIONS:
Overall Officials: ya x Xu, Principal Investigator — Zigong No.1 People's Hospital
Locations (1):
- Zigong First People's Hospital, Zigong, Sichuan, China